CLINICAL TRIAL: NCT02607254
Title: Efficacy and Safety of Pregabalin in Treatment of Neuropathic Pain in Patients With Idiopathic Small Fiber Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00054498
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Results first posted 2018-10-04 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Idiopathic Small Fiber Neuropathy
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin Treatment phase (Experimental): All patients will be initially treated with pregabalin in a single blind fashion
  Interventions: Drug: Pregabalin
- Withdrawal phase (Experimental): After finishing the treatment phase, some patients will be randomized to the placebo or continue on pregabalin for the 4 weeks of withdrawal phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Pregabalin will be given to the patients, starting at 75 mg BID and increased weekly to reach 225 mg BID for 8 weeks. During withdrawal phase, dose of pregabalin will be kept the same for patients who are randomized to the pregabalin withdrawal group.
  Other Names: Lyrica
  Arms: Pregabalin Treatment phase
Drug: Placebo — Placebo will be given to the patients that are randomized to placebo during withdrawal phase.
  Arms: Withdrawal phase

SUMMARY:
The purpose of this study is to assess safety and efficacy of treatment with pregabalin in patients with idiopathic small fiber neuropathy proven by skin biopsy.This is an enriched enrollment randomized withdrawal study that comprises 4 phases: a screening and selection phase, a washout period from previous pain medication for enriched enrollment, an 8 week single blind pregabalin treatment phase; and a 4 week randomized withdrawal phase.

DETAILED DESCRIPTION:
Patients who show any increase in their pain intensity score during the washout phase will be eligible for the single blind pregabalin treatment phase. Patients who respond to pregabalin, with at least 1 point improvement in neuropathic pain from baseline at the end of the single blind pregabalin treatment phase and meeting all other study requirements are considered eligible for participation in the withdrawal phase. These eligible patients are randomly assigned (1:1) to continue pregabalin or to be switched to placebo for a comparison of pregabalin efficacy and safety. Patients who have a worsening of average pain relative to the last week of the single blind pregabalin treatment period by more than one point and average pain level > =4 will be considered to have a loss of therapeutic response (LTR).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with idiopathic predominate-small fiber neuropathy
* Subject must have chronic peripheral neuropathic pain for more than 3 months
* A score >3 and <8 on Pain intensity scale for pain in prior week at first visit;
* Show increase in pain intensity scores during the wash off period;
* Age older than 18 years;

Exclusion Criteria:

* Subjects with large-fiber predominant neuropathy
* Subjects with HIV infection, trigeminal neuralgia (TGN), toxic neuropathy (e.g. chemotherapy exposure), paraneoplastic neuropathy, mono-gammopathy, inflammatory neuropathy, celiac disease, systemic lupus, peripheral vascular disease, connective tissue disorders, hepatitis C, Fabry disease, and diabetes;
* Subjects with uncontrolled thyroid or B12 disorders
* Subjects with Complex Regional Pain Syndrome
* Allergy to Pregabalin
* Subjects at risk of suicide or self harm
* Subjects with any clinically unstable cardiovascular, hematological, autoimmune, endocrine, renal, hepatic, renal, respiratory, or gastrointestinal disease; epilepsy, symptomatic peripheral vascular disease including intermittent claudication, pernicious anemia, untreated hypothyroidism, venous insufficiency, or spinal stenosis.
* History of known analgesic, alcohol or illicit drug abuse within 12 months of first visit;
* Pregnant females; breastfeeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-09; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Khoshnoodi, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11 subjects were recruited in the study.
Pre-assignment Details: Each subject underwent a washout period to stop the the current pain medications. Subjects who had significant reduction in pain were randomized to either placebo or Lyrica during the double blind withdrawal phase.
Groups:
- Pregabalin Treatment/Pregabalin Withdrawal: Patients in this arm were initially treated with pregabalin in a single blind fashion. After 8 weeks of treatment, they were randomized to continue on pregabalin for 4 weeks in the double blind randomized withdrawal phase as their pain was improved per protocol.
- Pregabalin Treatment/ Placebo Withdrawal: After finishing the pregabalin single-blinded treatment phase for 8 weeks, these patients were randomized to the placebo arm for the withdrawal phase for 4 weeks as their pain was improved during treatment phase.
- Pregabalin Treatment/No Withdrwal: These patients were treated with Pregabalin, but did not qualify for withdrawal phase as their pain did not improve to meet the criteria to enter the withdrawal phase.
Period: Overall Study
Arm/Group | Pregabalin Treatment/Pregabalin Withdrawal | Pregabalin Treatment/ Placebo Withdrawal | Pregabalin Treatment/No Withdrwal
Started | 3 | 3 | 5
Completed | 3 | 3 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pregabalin Treatment/Pregabalin Withdrawal: All patients will were with pregabalin. after 8 weeks of treatment, they were randomized to continue on pregabalin.
- Pregabalin Treatment/ Placebo Withdrawal: After finishing the pregabalin treatment phase for 8 weeks, these patients were randomized to the placebo arm for the withdrawal phase.
- Pregabalin Treatment/ No Withdrawal: After finishing the pregabalin treatment phase for 8 weeks, these patients did not qualify to continue to withdrawal phase.
- Total: Total of all reporting groups
Arm/Group | Pregabalin Treatment/Pregabalin Withdrawal | Pregabalin Treatment/ Placebo Withdrawal | Pregabalin Treatment/ No Withdrawal | Total
Number analyzed (Participants) | 3 | 3 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 5 | 11
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (6.4) | 47.3 (3.9) | 57.2 (7.1) | 53.4 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 7
  Male | 1 | 0 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 3 | 2 | 4 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Score for Pain Intensity.
Description: The primary outcome is change in visual analogue score for pain, with 0 being no pain at all and 10 being the most severe pain and a higher score meaning more pain, after 8 weeks of treatment phase and 4 weeks of randomized withdrawal phase.
Time Frame: Baseline, at 8 weeks after treatment phase and at 12 weeks for subjects completing the withdrawal phase
Population: Patient with idiopathic small fiber neuropathy.
Measure: Mean (Standard Deviation); unit: score on visual analogue score
Groups:
- Pregabalin Treatment/Pregabalin Withdrawal: All patients were initially treated with pregabalin. after 8 weeks of treatment, they were randomized to continue on pregabalin.
- Pregabalin Treatment/No Withdrwal: After finishing the 8 weeks pregabalin treatment phase, these patients did not qualify to enter the withdrawal phase.
Arm/Group | Pregabalin Treatment/Pregabalin Withdrawal | Pregabalin Treatment/ Placebo Withdrawal | Pregabalin Treatment/No Withdrwal
Number analyzed (Participants) | 3 | 3 | 5
score on visual analogue score
  Basline | 7.1 (1.4) | 6.9 (1.7) | 7.3 (2.3)
  After 8 weeks of Pregabalin | 5.4 (0.8) | 5.1 (1.1) | 7.6 (2.9)
  After 4 weeks of Withdrawal phase | 6.1 (1.2) | 7.4 (1.8) | NA (NA) — Patients did not qualify for the withdrawal phase.

2. Secondary Outcome: Brief Pain Inventory (BPI sf);
Description: Brief pain inventory is a scoring system for average pain intensity on scale of 0-10 with higher number meaning more pain.
Time Frame: Baseline, at 8 weeks after treatment phase and at 12 weeks for subjects completing the withdrawal phase
Population: Patients with idiopathic small fiber neuropathy.
Measure: Mean (Standard Deviation); unit: score in brief pain inventory scale
Groups:
- Pregabalin Treatment/Pregabalin Withdrawal: These patients were initially treated with pregabalin. after 8 weeks of treatment, they were randomized to continue on pregabalin if their pain is controlled.
- Pregabalin Treatment/ Placebo Withdrawal: After finishing the pregabalin treatment phase, these patients were randomized to the placebo arm for the withdrawal phase.
- Pregabalin Treatment/No Withdrwal: These patients did not qualify for the withdrawal phase after finishing the 8 weeks of pregabalin treatment.
Arm/Group | Pregabalin Treatment/Pregabalin Withdrawal | Pregabalin Treatment/ Placebo Withdrawal | Pregabalin Treatment/No Withdrwal
Number analyzed (Participants) | 3 | 3 | 5
score in brief pain inventory scale
  Basline | 6.7 (0.9) | 6.3 (1.1) | 7.2 (1.3)
  After 8 weeks of Pregabalin | 4.9 (1.1) | 4.5 (1.4) | 6.8 (1.7)
  After 4 weeks of Withdrawal phase | 5.8 (2.1) | 5.6 (1.9) | NA (NA) — These patients did not qualify for withdrawal phase.

3. Secondary Outcome: Sleep Quality as Assessed by Daily Sleep Interference Rating Scale (SIRS);
Description: a scoring system describing sleep quality between 0-10 with 0 having no problem with sleep and 10 not being to sleep at all.
Time Frame: Baseline, at 8 weeks after treatment phase and at 12 weeks for subjects completing the withdrawal phase
Population: Patients with idiopathic small fiber neuropathy
Measure: Mean (Standard Deviation); unit: score on Sleep Interference Rating scale
Groups:
- Pregabalin Treatment/Pregabalin Withdrawal: These patients were initially treated with pregabalin. After 8 weeks of treatment, They were randomized to continue on pregabalin.
- Pregabalin Treatment/ Placebo Withdrawal: After finishing the pregabalin treatment phase,these patients were randomized to the placebo arm for the withdrawal phase.
Arm/Group | Pregabalin Treatment/Pregabalin Withdrawal | Pregabalin Treatment/ Placebo Withdrawal | Pregabalin Treatment/No Withdrwal
Number analyzed (Participants) | 3 | 3 | 5
score on Sleep Interference Rating scale
  Basline | 4.5 (0.3) | 5.3 (0.61) | 5.9 (0.7)
  After 8 weeks of Pregabalin | 3.1 (0.65) | 2.8 (1.1) | 5.1 (1.5)
  After 4 weeks of Withdrawal phase | 3.9 (0.71) | 4.3 (0.87) | NA (NA) — These patients did not qualify for the withdrawal phase.

4. Secondary Outcome: Patient Global Impression of Change (PGIC);
Description: patient assign a number between 1-7 to the level of improvement, 1 showing substantial improvement and 7 showing no improvement at all.
Time Frame: At 8 weeks after treatment phase and at 12 weeks for subjects completing the withdrawal phase
Population: Patients with idiopathic small fiber neuropathy
Measure: Mean (Standard Deviation); unit: score on PGIC scale
Groups:
- Pregabalin Treatment/ Placebo Withdrawal: After finishing the 8 weeks of pregabalin treatment these patients were randomized to the placebo arm for the withdrawal phase.
Arm/Group | Pregabalin Treatment/Pregabalin Withdrawal | Pregabalin Treatment/ Placebo Withdrawal | Pregabalin Treatment/No Withdrwal
Number analyzed (Participants) | 3 | 3 | 5
score on PGIC scale
  After 8 weeks of pregabalin | 4.1 (0.31) | 5.4 (.61) | 1.8 (0.34)
  After Withdrawal phase | 3.9 (0.7) | 4.2 (1.11) | NA (NA) — These patients did not qualify for the withdrawal phase.

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Pregabalin Treatment/No Withdrawal: These patients were treated with Pregabalin, but did not qualify for withdrawal phase as their pain did not improve to meet the criteria to enter the withdrawal phase.
Arm/Group | Pregabalin Treatment/Pregabalin Withdrawal | Pregabalin Treatment/ Placebo Withdrawal | Pregabalin Treatment/No Withdrawal
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/5

LIMITATIONS AND CAVEATS:
There were low number of participants due to requirements of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT02607254/Prot_SAP_000.pdf